CLINICAL TRIAL: NCT07363213
Title: Assessment of Palatal Morphology and Age in Relation to Greater Palatine Canal/Foramen Anatomy on CBCT: A Retrospective Study in an Egyptian Population
Brief Title: Palatal Morphology, Age, and Greater Palatine Canal Anatomy on CBCT
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer of Periodontology, Department of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University., Cairo University
Other Study IDs: 12-2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Greater Palatine Foramen; Palatal Morphology
Keywords: greater palatine canal anatomy; palate morphology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to quantify the relationship between palatal morphology-including vault height, angle, width, and palatal bone thickness-and the dimensions and position of the greater palatine canal (GPC) and foramen (GPF). Secondary objectives include evaluating how age and sex relate to GPC/GPF measurements, as well as describing the prevalence and anatomical variations, including shapes, of accessory (lesser) palatine canals and foramina.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* CBCT scans showing complete hard palate
* Presence of first maxillary molars bilaterally

Exclusion Criteria:

* Palatal surgery or trauma history
* Maxillofacial anomalies
* Palatal pathology
* Poor CBCT quality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
the correlation between palatal morphology and the dimensions and position of the greater palatine canal (GPC) and foramen (GPF). | January 2026